CLINICAL TRIAL: NCT00001712
Title: Frequency of Parenteral and Non-Parenteral Exposures to Blood Among Healthcare Workers at the Clinical Center, NIH and at Seven Academic Hospitals in Japan
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980066; 98-CC-0066
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Hepatitis B; Hepatitis C; HIV Infection
Keywords: Healthcare Worker; Bloodborne Diseases; Hepatitis B; Hepatitis C; Human Immunodeficiency Virus; Parenteral Exposure; Non-Parenteral Exposure; Blood and Body Substances; Universal Precautions; HIV Seronegativity
MeSH Terms: conditions — Hepatitis B; Hepatitis C; HIV Infections; Acquired Immunodeficiency Syndrome

SUMMARY:
Following guidelines issued by the Centers for Disease Control, the Clinical Center implemented a Universal Precautions policy in November 1987 in an attempt to reduce healthcare workers' risks for occupational exposures to bloodborne pathogens. All hospital personnel whose jobs entailed potential exposure to patients' blood and body substances were required to attend a training session and complete a written examination. Based on data from surveys conducted before and twelve months after training in Universal Precautions, the frequency of cutaneous exposure to blood decreased by 50% in temporal association with implementation of Universal Precautions. Staff at the Clinical Center are required to take a refresher course in Universal Precautions annually.

The prevalence of bloodborne infections is high in Japan; however, Universal Precautions are not widely practiced in Japan. This study is designed: 1) to evaluate and compare nurses' knowledge of the epidemiology, pathogenesis, occupational risks, and appropriate prevention strategies for managing patients infected with bloodborne pathogens in the healthcare setting in seven university hospitals in Japan and at the Clinical Center of the National Institutes of Health in the US; 2) to compare self-reported levels of compliance with existing infection control recommendations designed to limit risk for exposure to bloodborne pathogens in all four institutions; 3) to compare self-reported frequencies of cutaneous exposures to blood at the four hospitals in the study; and 4) to evaluate the effect of educational intervention on nurses perceived compliance with recommendations and on the frequency of self-reported exposures to blood.

DETAILED DESCRIPTION:
Following guidelines issued by the Centers for Disease Control, the Clinical Center implemented a Universal Precautions policy in November 1987 in an attempt to reduce healthcare workers' risks for occupational exposures to bloodborne pathogens. All hospital personnel whose jobs entailed potential exposure to patients' blood and body substances were required to attend a training session and complete a written examination. Based on data from surveys conducted before and twelve months after training in Universal Precautions, the frequency of cutaneous exposure to blood decreased by 50% in temporal association with implementation of Universal Precautions. Staff at the Clinical Center are required to take a refresher course in Universal Precautions annually.

The prevalence of bloodborne infections is high in Japan; however, Universal Precautions are not widely practiced in Japan. This study is designed: 1) to evaluate and compare nurses' knowledge of the epidemiology, pathogenesis, occupational risks, and appropriate prevention strategies for managing patients infected with bloodborne pathogens in the healthcare setting in seven university hospitals in Japan and at the Clinical Center of the National Institutes of Health in the US; 2) to compare self-reported levels of compliance with existing infection control recommendations designed to limit risk for exposure to bloodborne pathogens in all four institutions; 3) to compare self-reported frequencies of cutaneous exposures to blood at the four hospitals in the study; and 4) to evaluate the effect of educational intervention on nurses perceived compliance with recommendations and on the frequency of self-reported exposures to blood.

ELIGIBILITY:
Nurses who work in the four cooperating institutions who have clinical responsibilities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3400
Dates: Start 1998-02; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fahey BJ, Koziol DE, Banks SM, Henderson DK. Frequency of nonparenteral occupational exposures to blood and body fluids before and after universal precautions training. Am J Med. 1991 Feb;90(2):145-53. PMID 1996583
- [Background] Willy ME, Dhillon GL, Loewen NL, Wesley RA, Henderson DK. Adverse exposures and universal precautions practices among a group of highly exposed health professionals. Infect Control Hosp Epidemiol. 1990 Jul;11(7):351-6. doi: 10.1086/646186. PMID 2376660
- [Background] Beekmann SE, Vlahov D, Koziol DE, McShalley ED, Schmitt JM, Henderson DK. Temporal association between implementation of universal precautions and a sustained, progressive decrease in percutaneous exposures to blood. Clin Infect Dis. 1994 Apr;18(4):562-9. doi: 10.1093/clinids/18.4.562. PMID 8038311